CLINICAL TRIAL: NCT03771248
Title: A Comparison Between Polyetheretherketone and Cobalt-chromium Telescopic Removable Partial Denture in Kennedy Class I Partially Edentulous Patients Regarding Oral Health Related Quality of Life (A Randomized Clinical Trial)
Brief Title: Polyetheretherketone vs Cobalt-chromium Telescopic Removable Partial Denture in Kennedy Class I Patients Regarding Oral Health Related Quality of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, tasneem gamal youssef el mashad, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Prosthesis1234
Record Dates: First submitted 2018-12-05; First posted 2018-12-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Partially Edentulous Mandible

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Co-cr telescopic partial denture (Active Comparator): A removable partial denture, that gains retention from a telescopic crown made of cobalt chromium
  Interventions: Device: peek telescopic partial denture
- PEEK telescopic partial denture (Experimental): A removable partial denture, its attachment is a telescopic crown made of PEEK
  Interventions: Device: peek telescopic partial denture

INTERVENTIONS:
Device: peek telescopic partial denture — removable partial denture

SUMMARY:
Dentistry is a rapidly progressing field with innumerable advances taking place on a day to day basis. The application of newer technologies and materials has advanced the specialty of prosthodontics and the services rendered to the patients.

Taking into consideration that PEEK as a material wasn't clinically investigated to be used as a material for routine use, however PEEK in removable partial dentures will help in making many steps easier and reach patients demands regarding esthetics. Also, owing to the superior mechanical and biological properties of PEEK, it will not be surprising if dentures constructed from the polymer are routinely constructed in near future.

DETAILED DESCRIPTION:
On fabrication of telescopic removable partial denture, choosing the material is a major step in the success of the treatment. There are different aspects that should be taken into consideration while choosing it. Beginning with retention as it is a crucial aspect. The retention of the telescopic partial denture is gained from the friction between the primary and secondary crowns. The chosen material should be able to maintain this type of retention for the longest possible period.

The esthetics also affects the treatment choice and patients preference, patients would choose metal free restorations over the ones that display metal. Finally the load distribution between the residual ridge and abutment should be equalized and transmitted in a favorable way. Otherwise one of the following consequences will occur; either overload on the abutment teeth followed by bone loss and abutment mobility or this overload is on the residual ridge leading to fast, progressive bone loss.

Cobalt chromium that is used for fabricating the telescopic removable partial denture is considered that most suitable material up till this moment. However, it doesn't fulfill much of the previous points.

As there will always be a continued improvement of materials and techniques used in dentistry especially in prosthodontics, innovative techniques must be regarded as potential alternatives to traditional materials.

PEEK is from the innovative materials that has shown promising results in different branches. However, to date no clinical studies or systematic reviews focusing on the use of PEEK dentures have been published, therefore more investigations are needed in this field.

ELIGIBILITY:
Inclusion Criteria:

* - Kennedy Class I Partially edentulous patients.
* Patients with good oral hygiene.
* The distal abutment bilaterally should be a premolar.
* Abutment teeth should be in a good periodontal condition.
* Sufficient inter-arch space, any super-eruptions should be treated before beginning of treatment.
* There should be no modifications spaces in the arch to be treated, and if found it should be treated with a fixed partial denture first.
* Normal tongue size
* Medically free from any disease that might affect bone support
* Patients with no history of bad oral habits as (Bruxism or Clenching) and free from any T.M.J disorders.

Exclusion Criteria:

* Patients with bad oral hygiene.
* Teeth with severe malalignment.
* The arch to be treated is opposed by a completely edentulous arch.
* Unmotivated patient.
* Patient with a medical disease that will hinder his ability to be committed to the treatment.
* Patients on a radiation therapy.
* Patients with xerostomia.
* Patients with a history of drug, alcohol abuse or psychiatric disorder.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
oral health impact profile | 12 months
  questionnaire

SECONDARY OUTCOMES:
probing depth of abutment teeth | 12 months
  using williams graduated probe
abutment mobility | 12 months
  millers classification